CLINICAL TRIAL: NCT04425993
Title: Rectal Indomethacin Versus Rectal Indomethacin and Sublingual Nitrate to Prevent Post-ERCP Pancreatitis: a Multicentre, Non-inferiority, Double-blind, Randomised Trial
Brief Title: Rectal Indomethacin Versus Rectal Indomethacin and Sublingual Nitrate for PEP Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20200522-4
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: ERCP; Post-ERCP pancreatitis; PEP; NSAIDs; indomethacin; nitrate
MeSH Terms: interventions — Isosorbide Dinitrate; Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rectal indomethacin and sublingual nitrate (Experimental): All patients without contraindications should receive sublingual isosorbide dinitrate within 5 min before ERCP.
  All patients without contraindications should receive rectal indomethacin within 30 min before ERCP.
  Interventions: Drug: Isosorbide Dinitrate 5 MG; Drug: Indomethacin 100 MG
- Rectal indomethacin and sublingual placebo (Active Comparator): All patients without contraindications should receive sublingual placebo within 5 min before ERCP.
  All patients without contraindications should receive rectal indomethacin within 30 min before ERCP.
  Interventions: Drug: Indomethacin 100 MG; Drug: Sublingual Placebo
- Rectal placebo and sublingual nitrate (Active Comparator): All patients without contraindications should receive sublingual isosorbide dinitrate within 5 min before ERCP.
  All patients without contraindications should receive rectal placebo within 30 min before ERCP.
  Interventions: Drug: Isosorbide Dinitrate 5 MG; Drug: Rectal placebo
- Rectal placebo and sublingual placebo (Placebo Comparator): All patients without contraindications should receive sublingual placebo within 5 min before ERCP.
  All patients without contraindications should receive rectal placebo within 30 min before ERCP.
  Interventions: Drug: Sublingual Placebo; Drug: Rectal placebo

INTERVENTIONS:
Drug: Isosorbide Dinitrate 5 MG — All patients without contraindications should receive sublingual isosorbide dinitrate tablet within 5 minutes before ERCP.
  Arms: Rectal indomethacin and sublingual nitrate; Rectal placebo and sublingual nitrate
Drug: Indomethacin 100 MG — All patients without contraindications should receive rectal indomethacin within 30 min before ERCP.
  Arms: Rectal indomethacin and sublingual nitrate; Rectal indomethacin and sublingual placebo
Drug: Sublingual Placebo — All patients without contraindications should receive sublingual placebo within 5 minutes before ERCP.
  Arms: Rectal indomethacin and sublingual placebo; Rectal placebo and sublingual placebo
Drug: Rectal placebo — All patients without contraindications should receive rectal placebo within 30 min before ERCP.
  Arms: Rectal placebo and sublingual nitrate; Rectal placebo and sublingual placebo

SUMMARY:
Patients undergoing endoscopic retrograde cholangiopancreatography (ERCP) are at risk for post-ERCP pancreatitis (PEP), which is associated with adverse outcomes. Combination prophylaxis strategies are increasingly investigated to prevent PEP more effectively, and studies have confirmed the benefits. Two randomized controlled trials revealed that combination prophylaxis with rectal NSAIDs and sublingual nitrate has reduced PEP rates to 5.6%-6.7% in average-risk patients. However, there was concern regarding the safety of sublingual nitrate with reports of significant increasing the risk of hypotesion (rate of 54.9%) and headache (rate of 4.1%) as compared with placebo.

As a safety drug, rectal administration of one dose NSAIDs is recommended as basic chemoprophylaxis in common or high-risk patients in guidelines. Results from previous studies showed rectal administration of NSAIDs significantly reduced PEP rate to 4-5.3% in average-risk patients. Although the difference in demographics, study design and outcomes definition, evidence was obtained that rectal NSAIDS was associated with similar PEP rate as combination prophylaxis with rectal NSAIDs and sublingual nitrate. However, evidence is lacking from large, randomized clinical trials indicating that efficiency of PEP prevention with rectal NSAIDs alone is not inferior to with combination prophylaxis. The investigators conduct this trial to investigate the hypothesis that rectal NSAIDs alone is non-inferior to the combination prophylaxis in terms of PEP prevention, but with reduce side effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age, 18-80 y) with native papilla planned for diagnostic or therapeutic ERCP were eligible for enrollment in the study.

Exclusion Criteria:

* contraindications to ERCP;
* allergy to nitrates or NSAIDs;
* currently on nitrate medication;
* receiving NSAIDs within 7 days;
* not suitable for indomethacin eg, gastrointestinal hemorrhage within the past 4 weeks, renal dysfunction (creatinine level >1.4 mg/dL) or the presence of coagulopathy before the procedure (international normalized ratio > 1.5);
* acute pancreatitis within 3 days;
* pregnant or breastfeeding women;
* unwilling or inability to provide consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of post-ERCP Pancreatitis | 14 days
  The diagnosis of PEP was established if there was new onset of upper abdominal pain associated with an increased amylase or lipase level of at least 3 times the upper limit of normal range at 24 hours after the procedure, and hospitalization for at least 2 nights. Doctors are advised to use cross-sectional imaging to identify ambiguous PEP.

SECONDARY OUTCOMES:
Rate of moderate to severe PEP | 14 days
  The severity classification of pancreatitis was defined according to the criteria of Cotton et al and the revised Atlanta criteria.
Other adverse events | 14 days
  Adverse effects of indomethacin, including gastrointestinal bleeding and renal failure.
  Adverse effects of nitrates, including hypotension, headache and dizziness. Other post-ERCP adverse events including cholangitis, bleeding, and perforation.
  Any other adverse outcomes possibly related to ERCP or experimental drugs that required hospital admission or a prolonged hospital stay for further management.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Xiamen Humanity Hospital, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xijing Hoapital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sotoudehmanesh R, Eloubeidi MA, Asgari AA, Farsinejad M, Khatibian M. A randomized trial of rectal indomethacin and sublingual nitrates to prevent post-ERCP pancreatitis. Am J Gastroenterol. 2014 Jun;109(6):903-9. doi: 10.1038/ajg.2014.9. Epub 2014 Feb 11. PMID 24513806
- [Background] Tomoda T, Kato H, Ueki T, Akimoto Y, Hata H, Fujii M, Harada R, Ogawa T, Wato M, Takatani M, Matsubara M, Kawai Y, Okada H. Combination of Diclofenac and Sublingual Nitrates Is Superior to Diclofenac Alone in Preventing Pancreatitis After Endoscopic Retrograde Cholangiopancreatography. Gastroenterology. 2019 May;156(6):1753-1760.e1. doi: 10.1053/j.gastro.2019.01.267. Epub 2019 Feb 14. PMID 30772342
- [Background] Ding J, Jin X, Pan Y, Liu S, Li Y. Glyceryl trinitrate for prevention of post-ERCP pancreatitis and improve the rate of cannulation: a meta-analysis of prospective, randomized, controlled trials. PLoS One. 2013 Oct 1;8(10):e75645. doi: 10.1371/journal.pone.0075645. eCollection 2013. PMID 24098392
- [Background] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971
- [Background] Luo H, Wang X, Zhang R, Liang S, Kang X, Zhang X, Lou Q, Xiong K, Yang J, Si L, Liu W, Liu Y, Zhou Y, Wang S, Yang M, Chen W, Han Y, Shang G, Yang X, He Y, Zou Q, Guo W, Dai Y, Zeng W, Zhu X, Gong R, Li X, Nie Z, Wang Q, Wang L, Pan Y, Guo X, Fan D. Rectal Indomethacin and Spraying of Duodenal Papilla With Epinephrine Increases Risk of Pancreatitis Following Endoscopic Retrograde Cholangiopancreatography. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1597-1606.e5. doi: 10.1016/j.cgh.2018.10.043. Epub 2018 Oct 31. PMID 30391434